CLINICAL TRIAL: NCT01365780
Title: Identification of Microcirculation in Distal Radius Fractures After Surgical Treatment With and Without Hyperbaric Oxygen Therapy (HBOT)
Brief Title: Hyperbaric Oxygen Therapy in Distal Radius Fractures: Can it Shorten Recovery Time and Increase Fracture Healing?
Acronym: HBOTRadius
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: nump
  acceptence by patient too low
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTC-A10-29
Record Dates: First submitted 2011-06-01; First posted 2011-06-03 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Hyperbaric Oxygen Therapy; Recovery Time; Contrast Media; Sonography
Keywords: microcirculation, O2c
MeSH Terms: interventions — Hyperbaric Oxygenation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- With HBOT (Active Comparator): Patients, who receive hyperbaric Oxygen Therapy after their surgical treatment
  Interventions: Procedure: Hyperbaric Oxygen Therapy
- Without HBOT (No Intervention): Patients who receive the same surgical treatment of their radius fracture than the patients of the group "with HBOT", but no hyperbaric oxygen therapy (comparison group)

INTERVENTIONS:
Procedure: Hyperbaric Oxygen Therapy — The patients receive 10 sessions of HBOT in two weeks, starting on the day after the surgical treatment of their radius fracture. Each session lasts about one hour.
  Arms: With HBOT

SUMMARY:
This project is meant to show wether the HBOT can fasten the recovery process after surgical treatment of distal Radius fractures. For this propose the microcirculation is measured, together with the level of pain on a visual analog scale (VAS) and the remaining force of the hand after surgery is examined. Furthermore the sonography with contrast medium which is long established for examination of organs of the parenchyma, is meant to be verified at the muscular-skeletal system in this project.

DETAILED DESCRIPTION:
This project investigates microcirculation in skin, muscle and bone after surgical treatment of distal Radius fracture with and without Hyperbaric Oxygen Therapy for detecting any benefit of the HBOT. In Hyperbaric Oxygen Therapy the patients breathes Oxygen from a mask in a pressure chamber with higher air pressure than normal atmospheric pressure wich is meant to increase the peripheric oxygen suppley in the healing tissue. The patients will receive 10 sessions of HBOT. The patients who are treated with HBOT are chosen randomly.

The microcirculation is measured as parameter for tissue damage and wound healing. It is registered by O2c, which works with measuring reflected lightwaves. It is strictly noninvasive and causes absolutely no pain for the patient. The measurement device consists of two small probes, which simply stick to the patient´s skin. There are 8 measurements in this study:

The first one shortly after the surgical treatment, then there will be one measuring appointment every week up to four week. Afterwards the patients hands will be measured in the 6th, 8th and 12th week after surgical treatment. In all measurements the healthy side will be measured as well for comparison. Additional the force fo both hands and the level of pain in the Visual Analogue Scale are evaluated.

Furthermore there will be a sonography with contrast medium in the first week after surgical treatment to indicate any increase of blood suppley after the HBOT and detect any wound healing complications.

Therefore this study will research on the one hand if there is a benefit to the HBOT for the often young and healthy patients of radius fractures to return earlier and more easily to their health condition. On the other hand this study is meant to establish the sonography with contrast medium as a examination method with little risks.

ELIGIBILITY:
Inclusion Criteria:

* distal radius fracture
* only one radius is fractured
* medical treatment within 72 hours after accident
* patient will receive surgical treatment (plate)
* patient received information letter and singed agreement
* patient is German-speaking
* patient is competent
* patient is over 18 years of age

Exclusion Criteria:

* pathologic fractures
* open fractures
* fractures with wide soft tissue damage, that affects surgical treatment
* surgical treatment after more than 72 hours after the accident
* diabetes mellitus, that need medical treatment
* patient has PAD
* previous surgery treatment on the fractured arm or refracture
* patient is not competent
* immune deficiency
* polytrauma
* patient with diseases of the lung (hypercapnia)
* patient with open Foramen ovale
* pregnant women
* patient with NYHA IV

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2011-09; Primary Completion 2012-11 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
functional outcome | 18 months
  The functional outcome is measured by microcirculation as parameter for wound healing, force of the treated hand and level of pain.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Knobe, MD, Principal Investigator — Dpt. of Orthopedic Trauma, RWTH Aachen University; Hans-Christoph Pape, Univ.-Prof. MD FACS, Study Chair — Dpt. of Orthopedic Trauma, RWTH Aachen University
Locations (1):
- RWTH Aachen University Hospital, Aachen, North Rhine-Westphalia, Germany